CLINICAL TRIAL: NCT01236261
Title: Prospective Population Study on Candidemia in Spain (Estudio Poblacional Prospectivo Sobre Candidemia en España)
Brief Title: Prospective Population Study on Candidemia in Spain
Acronym: CANDIPOP
Status: Completed | Type: Observational
Sponsor: Fundacion SEIMC-GESIDA (Other)
Collaborators: Astellas Pharma Inc (Industry); Gilead Sciences (Industry); Merck Sharp & Dohme LLC (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: GEMICOMED-GEIH 0109
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Fungemia
Keywords: Fungemia, fungal infection, susceptibility, antifungal
MeSH Terms: conditions — Fungemia; Mycoses; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fungal strains obtained from blood cultures.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fungemia: Patients with a fungal isolate from a blood culture
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — Non interventional study

SUMMARY:
The aim of this study is to describe the epidemiology of fungal blood infections in Spain (with emphasis on the incidence, fungal species distribution and antifungal susceptibility). The study is to be performed in five big cities which represent different geographic areas: Barcelona, Bilbao, Madrid, Sevilla and Valencia.

ELIGIBILITY:
Inclusion Criteria:

* Fungal isolate obtained from blood sample

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Candida sp or other fungal isolate obtained from a blood sample (fungemia episode)
Sampling Method: Non-Probability Sample
Enrollment: 730 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Describe fungemia epidemiology in Spain | 1 year
  Recollection of demographic variables (age, gender and ethnic origin); clinical variables (background diseases, other coinfections, treatment received, etc) and microbiological information of the isolate.

SECONDARY OUTCOMES:
Describe differences among cities and institutions | 1 year
  Analyze results in function of the city and hospital where the isolate was obtained (5 cities in Spain and 29 participating hospitals)
Definition of risk factors | 1 year
  Determine risk factors for:
  * bad clinical evolution
  * infection by a specific Candida species
  * fluconazole resistant isolate
  * fungemia persistency
Determination of the fungal isolates susceptibility to fluconazole, voriconazole, caspofungine, anidulafungine, micafungine and anfotericine B | 1 year
  Analysis of resistant strains percentage according to the threshold established by CLSI to each specific antifungal
Correlation between fungemia with a diminished susceptibility fungal strain and clinical evolution | 1 year
  Chi-square and Kaplan-Meier survival curves
Correlation between reference and commercial microbiological methods | 1 year
  Comparison of results when a reference or a commercial fungal identification and antifungal susceptibility method is used.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Cuenca, MD, PhD, Study Director — Instituto de Salud Carlos III; Belen Padilla, MD, Study Director — Hospital Gregorio Marañon; Isabel Ruiz, MD, Study Director — Hospital Vall d'Hebron; Jose Garnacho-Montero, MD, Study Director — Hospital Virgen del Rocio
Locations (29):
- Spain (29):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital de Barcelona, Barcelona, Barcelona
  - Hospital Vall d'Hebrón, Barcelona, Barcelona
  - Hospital Clinic i Provincial, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Sant Joan de Dèu, Esplugues de Llobregat, Barcelona
  - Hospital Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital de la Princesa, Madrid, Madrid
  - Hospital Gregorio Marañon, Madrid, Madrid
  - Hospital del Niño Jesús, Madrid, Madrid
  - Hospital Infanta Leonor, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital 12 de Octubre, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital San Juan de Dios del Aljarafe, Bormujos, Seville
  - Hospital Virgen de Macarena, Seville, Seville
  - Clínica Sagrado Corazón, Seville, Seville
  - Hospital Virgen del Rocío, Seville, Seville
  - Hospital Nuestra Señora de Valme, Seville, Seville
  - Hospital La Fe, Valencia, Valencia
  - Hospital Clínico de Valencia, Valencia, Valencia
  - Hospital General de Valencia, Valencia, Valencia
  - Hospital Doctor Peset, Valencia, Valencia
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital de Basurto, Basurto, Vizcaya
  - Hospital de Galdakao-Usansolo, Galdakao, Vizcaya

REFERENCES:
- [Derived] Puig-Asensio M, Fernandez-Ruiz M, Aguado JM, Merino P, Lora-Pablos D, Guinea J, Martin-Davila P, Cuenca-Estrella M, Almirante B. Propensity Score Analysis of the Role of Initial Antifungal Therapy in the Outcome of Candida glabrata Bloodstream Infections. Antimicrob Agents Chemother. 2016 May 23;60(6):3291-300. doi: 10.1128/AAC.00195-16. Print 2016 Jun. PMID 26976872